CLINICAL TRIAL: NCT06994637
Title: Effects of Liquid Hourglass and Spiky Ball on Pain, Fear, Anxiety and Emotional Manifestations During Venous Blood Collection in Children: A Randomized Controlled Study
Brief Title: Effects of Liquid Hourglass and Spiky Ball on Pain, Fear, Anxiety and Emotional Manifestations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hakkari Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Demir Kösem, Assistant Professor, Hakkari Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HakkariU
Record Dates: First submitted 2025-04-26; First posted 2025-05-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pain; Anxiety and Fear; Procedural Anxiety; Procedural Pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Intervention Group-Liquid Hourglass Group: The liquid hourglass method will be applied to the children in this group as a non-pharmacological application. Children will be given a liquid hourglass and during the blood collection process, the researcher or parent will turn it and watch the colored bubbles made by the liquid gel flow down by drop, and they will be allowed to take the liquid hourglass with their free hand if they wish.
  Intervention Group-Spiky Ball Group: The children in this group will be applied the spiky ball method as a non-pharmacological application. Children will be given a spiky ball and asked to hold the ball in the palm of the arm where the blood collection process is performed.
  Control Group: The child will be seated in the intervention chair. No pharmacological or non-pharmacological method will be applied to the children in this group other than the routine blood collection process.
Who Masked: Outcomes Assessor
Masking Description: To minimize potential bias during data collection, all assessments were conducted by an independent nurse who was not involved in the study. However, due to the visible and interactive nature of the interventions, blinding of participants, parents, and the nurse performing the procedure was not feasible. To prevent allocation bias, the randomization table was created by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liquid Hourglass (Experimental): Liquid Hourglass: The liquid hourglass to be used in the study is approximately 14 cm long and made of high-quality plastic material. It contains colored liquid gel. When the hourglass is turned, the colored liquid gel inside flows downwards in the form of bubbles, drop by drop. It is suitable for use by all age groups of children.
  The liquid hourglass method will be applied to the children in this group as a non-pharmacological application. Children will be given a liquid hourglass and during the blood collection process, the researcher or parent will turn it and watch the colored bubbles made by the liquid gel flow down by drop, and they will be allowed to take the liquid hourglass with their free hand if they wish. The liquid hourglass will be cleaned with alcohol after it is used on each child. The blood collection process will be performed by the nurse working in the blood collection unit.
  Interventions: Other: Liquid Hourglass
- Spiky Ball (Experimental): Spiky Ball: The spiky ball to be used in the study is a ball made of sturdy environmentally friendly plastic, approximately 6 cm in size. This ball has a hard body with thorns on it and provides tactile stimulation by pricking the child's fingers. The pressure applied by the thorns on the balls to the hand can reduce pain, muscle tension and stress by stimulating the nerve endings more quickly. It is suitable for use by children over the age of two. The tactile stimulation on the spiky ball can distract the child during the blood collection process.
  The children in this group will be applied the spiky ball method as a non-pharmacological application. Children will be given a spiky ball and asked to hold the ball in the palm of the arm where the blood collection process is performed. The spiky ball will be cleaned with alcohol after it is used on each child. The blood collection process will be performed by the nurse working in the blood collection unit.
  Interventions: Other: Spiky Ball
- Control Group (No Intervention): The child will be seated in the intervention chair. No pharmacological or non-pharmacological method will be applied to the children in this group other than the routine blood collection process. The blood collection process will be performed by the nurse working in the blood collection unit.

INTERVENTIONS:
Other: Liquid Hourglass — The liquid hourglass to be used in the study is made of high-quality plastic material, approximately 14 cm long. It contains colored liquid gel. When the hourglass is turned, the colored liquid gel inside flows downwards in the form of bubbles, drop by drop. It is suitable for use by all age groups of children. The visual and moving nature of the liquid hourglass may distract the child during the blood collection process.
  Arms: Liquid Hourglass
Other: Spiky Ball — The spiky ball to be used in the study is a ball made of sturdy environmentally friendly plastic, approximately 6 cm in size. This ball has a hard body with thorns on it and provides tactile stimulation by pricking the child's fingers. The pressure applied by the thorns on the balls to the hand can reduce pain, muscle tension and stress by stimulating the nerve endings more quickly. It is suitable for use by children over the age of two. The tactile stimulation on the spiky ball can distract the child during the blood collection process.
  Arms: Spiky Ball

SUMMARY:
This research will be conducted as a pre-test-post-test parallel group randomized controlled experimental study to determine the effects of liquid hourglass and spiky ball applied during venous blood collection on pain, fear, anxiety and emotional indicators in children aged 4-6.

Research Hypotheses H1: The mean pain scores of children in the liquid hourglass group are lower than the mean scores of children in the control group.

H2: The mean fear scores of children in the liquid hourglass group are lower than the mean scores of children in the control group.

H3: The mean anxiety scores of children in the liquid hourglass rod group are lower than the mean scores of children in the control group.

H4: The mean emotional indicator scores of children in the liquid hourglass rod group are lower than the mean scores of children in the control group.

H5: The mean pain scores of children in the spiky ball group are lower than the mean scores of children in the control group.

H6: The mean fear scores of children in the spiky ball group are lower than the mean scores of children in the control group.

H7: The mean anxiety scores of children in the spiky ball group are lower than the mean scores of children in the control group.

H8: The mean emotional indicator scores of children in the spiky ball group are lower than the mean scores of children in the control group.

DETAILED DESCRIPTION:
The most common invasive procedures that children encounter, such as blood collection, peripheral vascular access, injection, and lumbar puncture, are among the painful and disturbing procedures. These procedures can cause pain, fear, and anxiety in children. Especially between the ages of three and six, children have magical thoughts about the disease due to their immature abstract thinking and cause-effect skills, and may perceive pain, fear, and painful situations as punishment for not listening to their parents. Considering these developmental characteristics of preschool children, it is important to make the process less stressful with appropriate support and guidance during painful medical procedures and to better respond to children's emotional needs. In particular, blood collection is among the medical interventions in which these emotional reactions are experienced most intensely. Unmanaged pain, fear, and anxiety related to these procedures in children can cause many physiological and psychological consequences. These negative experiences can lead to maladaptive pain reactions, poor cognitive and motor development, needle phobia, avoidance of healthcare personnel and services, and long-term traumatic memories that can continue throughout adulthood. For these reasons, managing pain, anxiety, and fear in children is very important. Management of pain, anxiety, and fear requires a multidisciplinary team to work collaboratively. The nurse has an indispensable role in this team. The American Association of Pain Management Nursing reported that nurses are responsible for providing pain control using pharmacological and non-pharmacological methods before, during, and after interventions in individuals exposed to painful procedures. Non-pharmacological methods that can be used in the effective management of pain are among the independent care roles of nurses. Non-pharmacological methods are classified as physical, cognitive-behavioral, and other supportive methods. Distraction intervention, one of the cognitive-behavioral methods, aims to alleviate pain, stress, and anxiety during painful procedures in pediatric patients by directing attention from a painful stimulus to an interesting object or a non-threatening, pleasant stimulus. Among these, applications such as watching cartoons or videos, distraction cards, virtual reality, blowing balloons and coughing, listening to music, playing games, and using a kaleidoscope support the reduction of pain, fear, and anxiety by diverting attention from painful stimuli. Among the physical methods, Buzzy, ShotBlocker, hot or cold applications, massage, providing stimulation to the skin, and giving a ball to the palm are the methods used to reduce pain, anxiety, and fear. Nowadays, in addition to the products available on the market to reduce pain and anxiety, there is an increasing interest in innovative methods. Based on this, in the scope of the research we planned, unlike previous studies, we wanted to examine the liquid hourglass and spiky ball.

One of the attention-grabbing methods used for pain, fear and anxiety management in medical procedures in children may be the liquid hourglass method. It is a cheap, easy, effective, side-effect-free and safe intervention to help children cope. It is stated that the liquid moving hourglass can be successful in distracting pediatric patients because the colored bubbles provide a calming and visually stimulating experience while floating and descending. Studies have shown that visual and moving toys reduce children's pain, fear and anxiety levels during the blood collection procedure. When the literature is examined, no study has been found examining the effect of liquid hourglass applied during blood collection on pain, fear and anxiety in children. Distraction methods are supported by various tactile stimulation tools. Tactile stimulation distracts the child's attention and focuses his/her attention away from painful sensations and on tactile stimulation, thus reducing the sensation of pain. Tactile stimulation is frequently used for the management of pain in invasive procedures. Tactile stimulation is an intervention that has the potential to block pain transmission. According to the gate control theory, tactile stimulation produced by physical interventions closes the pain gate in the spinal cord and helps reduce the level of pain by increasing the activation of somatosensory sensory areas. In addition, since the stimuli cross the spinal cord, the tactile stimulus can be applied directly to the painful area, proximal or distal to that area, and symmetrically opposite (contralateral) to the painful area. The spiky ball application is designed as a plastic apparatus with a hard body with thorny protrusions that generate tactile stimulation from the palm. The pressure applied by the thorns on the balls to the hand stimulates the nerve endings more quickly, which can reduce the pain, muscle tension, and stress experienced by children during invasive procedures. It has been determined that there are limited studies in the literature using a spiky ball as a tactile stimulus from the palm to reduce pain, fear and anxiety during venous blood sampling.

Since there are no studies examining the effect of using liquid hourglass on reducing pain, fear and anxiety during blood collection in children and the use of spiky balls is limited, it is thought that the study will add new information to the literature and contribute to reducing the problems caused by painful applications for children, their families and pediatric nurses with the use of new methods.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 4-6 years old
* The child and parent must agree to participate in the research
* The child and parent must be able to speak Turkish

Exclusion Criteria:

* The child is not in the appropriate age range
* The child is in pain
* The child has a mental or auditory disability
* The child is unconscious
* The child and parent do not agree to participate in the study

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Pain During Venous Blood Collection in Children | "2 months"
  "Pain is a specific unpleasant sensation originating from any part of the body, encompassing all past experiences of a person, whether or not due to an organic cause."

OTHER OUTCOMES:
Fear During Venous Blood Collection in Children | "2 months"
  "It is a vital response that occurs as a response to a stimulus that is perceived as a specific pain or threat."
Anxiety During Venous Blood Collection in Children | "2 months "
  "It is a common psychological disorder that causes a person to have excessive and uncontrollable reactions to emotions such as worry, anxiety and fear."
Emotional Manifestation During Venous Blood Collection in Children | "2 months "
  "It is the name given to the emotional states of people."

CONTACTS AND LOCATIONS:
Locations (1):
- Hakkari University, Hakkâri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No